CLINICAL TRIAL: NCT05096208
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF 3 LOTS OF RESPIRATORY SYNCYTIAL VIRUS (RSV) PREFUSION F SUBUNIT VACCINE IN HEALTHY ADULTS
Brief Title: Clinical Lot Consistency for RSVpreF in a Population of Healthy Adults 18 to ≤49 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C3671014
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: RSV
Keywords: RSV; Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded, placebo controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RSVpreF vaccine Group 1 (Experimental): RSVpreF
  Interventions: Biological: RSVpreF (Group 1)
- RSVpreF vaccine Group 2 (Experimental): RSVpreF
  Interventions: Biological: RSVpreF (Group 2)
- RSVpreF vaccine Group 3 (Experimental): RSVpreF
  Interventions: Biological: RSVpreF (Group 3)
- Placebo dose (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSVpreF (Group 1) — RSV vaccine (RSVpreF)
  Arms: RSVpreF vaccine Group 1
Biological: RSVpreF (Group 2) — RSV vaccine (RSVpreF)
  Arms: RSVpreF vaccine Group 2
Biological: RSVpreF (Group 3) — RSV vaccine (RSVpreF)
  Arms: RSVpreF vaccine Group 3
Biological: Placebo — Placebo
  Arms: Placebo dose

SUMMARY:
This randomized, double-blinded, placebo-controlled Phase 3 study is designed to evaluate the safety, tolerability, and immunogenicity of 3 lots of RSVpreF in healthy adults.

DETAILED DESCRIPTION:
This randomized, double-blinded, placebo-controlled Phase 3 study will examine the immune response and the safety and tolerability profiles across 3 manufactured lots of RSVpreF when administered as a single 120 µg dose to healthy adults to demonstrate lot equivalence in manufacturing of RSVpreF.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or nonpregnant, nonbreastfeeding females between the ages of 18 and ≤49 years, inclusive, at Visit 1 (Day 1).
2. Participants who are willing and able to comply with scheduled visits, laboratory tests, lifestyle considerations, and other study procedures, including daily completion of the e diary for 7 days after study vaccination.
3. Healthy participants as determined by medical history, physical examination (if required), and the clinical judgment of the investigator to be eligible for inclusion in the study. Participants with preexisting chronic medical conditions determined to be stable in the clinical judgment of the investigator may be included.
4. Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the ICD and in the protocol.

Exclusion Criteria:

1. Bleeding diathesis or condition associated with prolonged bleeding time that may contraindicate IM injection.
2. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention or any related vaccine.
3. Unstable chronic medical condition or disease requiring significant change in therapy or hospitalization for worsening disease within 3 months before receipt of study intervention.
4. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
5. Known infection with HIV, HCV, or HBV.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
7. Previous vaccination with any licensed or investigational RSV vaccine at any time prior to enrollment or planned receipt throughout the study.
8. Receipt of any blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
9. Receipt of monoclonal antibodies from 60 days before study intervention administration or planned receipt throughout the study.
10. Receipt of systemic treatment with known immunosuppressant medications within 60 days before study intervention administration or the use of systemic corticosteroids (≥20 mg/day of prednisone or equivalent) for ≥14 days within 28 days prior to study enrollment. Prednisone use of <20 mg/day for <14 days is permitted. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin, eyes, ears) corticosteroids are permitted.
11. Current alcohol abuse or illicit drug use. Note: Marijuana use is not considered an exclusion criterion for the study when elicited in participant screening, though it may be considered illicit in some locales.
12. Current use of any prohibited concomitant medication(s) or those unwilling/unable to use a permitted concomitant medication(s).
13. Participation in other studies involving investigational drug(s) or investigational vaccines within 28 days prior to consent and/or during study participation.
14. Pregnant females; breastfeeding females; and women of child bearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in the protocol for the duration of the study.
15. Men who are unwilling to comply with contraception methods as outlined in the protocol for the duration of the study.
16. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1028 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Clinical Site Partners, Inc, Winter Park, Florida
  - Clinical Site Partners, Winter Park, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Clinical Research Prime, Idaho Falls, Idaho
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Aventiv Research Inc, Columbus, Ohio
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Benchmark Research, Austin, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Baker J, Aliabadi N, Munjal I, Jiang Q, Feng Y, Brock LG, Cooper D, Anderson AS, Swanson KA, Gruber WC, Gurtman A. Equivalent immunogenicity across three RSVpreF vaccine lots in healthy adults 18-49 years of age: Results of a randomized phase 3 study. Vaccine. 2024 May 10;42(13):3172-3179. doi: 10.1016/j.vaccine.2024.03.070. Epub 2024 Apr 16. PMID 38616438
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671014

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1028 participants signed the informed consent form (ICF) and were enrolled. Out of which, 35 participants were not eligible for randomization and 993 participants were randomized into the study. Only 992 participants were vaccinated.
Groups:
- Placebo: Participants were randomized to receive a single intramuscular injection of placebo reconstituted with sterile water for injection, once only on Day 1.
- Group 1: RSVpreF Lot 1: Participants were randomized to receive a single intramuscular injection of 120 microgram (mcg) Respiratory Syncytial Virus prefusion F subunit vaccine (RSVpreF) Lot 1 reconstituted with sterile water for injection, once only on Day 1.
- Group 2: RSVpreF Lot 2: Participants were randomized to receive a single intramuscular injection of 120 mcg RSVpreF Lot 2 reconstituted with sterile water for injection, once only on Day 1.
- Group 3: RSVpreF Lot 3: Participants were randomized to receive a single intramuscular injection of 120 mcg RSVpreF Lot 3 reconstituted with sterile water for injection, once only on Day 1.
Period: Overall Study
Arm/Group | Placebo | Group 1: RSVpreF Lot 1 | Group 2: RSVpreF Lot 2 | Group 3: RSVpreF Lot 3
Started | 247 | 249 | 247 | 250
Vaccinated | 247 | 249 | 247 | 249
Completed | 243 | 243 | 239 | 245
Not Completed | 4 | 6 | 8 | 5
Not completed — Lost to Follow-up | 3 | 5 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 3
Not completed — No longer met eligibility criteria | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received study intervention.
Groups:
- Group 1: RSVpreF Lot 1: Participants were randomized to receive a single intramuscular injection of 120 mcg RSVpreF Lot 1 reconstituted with sterile water for injection, once only on Day 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Group 1: RSVpreF Lot 1 | Group 2: RSVpreF Lot 2 | Group 3: RSVpreF Lot 3 | Total
Number analyzed (Participants) | 247 | 249 | 247 | 249 | 992
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.46 (8.73) | 34.16 (8.58) | 33.81 (9.02) | 33.90 (9.02) | 34.08 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 138 | 158 | 157 | 593
  Male | 107 | 111 | 89 | 92 | 399
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 65 | 68 | 55 | 248
  Not Hispanic or Latino | 185 | 180 | 174 | 189 | 728
  Unknown or Not Reported | 2 | 4 | 5 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 2 | 8
  Asian | 6 | 16 | 7 | 9 | 38
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 4 | 6
  Black or African American | 48 | 53 | 53 | 50 | 204
  White | 178 | 169 | 177 | 179 | 703
  More than one race | 7 | 4 | 5 | 1 | 17
  Unknown or Not Reported | 5 | 5 | 2 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratios (GMRs) of Respiratory Syncytial Virus Subgroup A (RSV A) and B (RSV B) Neutralizing Antibodies at 1 Month After Vaccination for Every Pair of RSVpreF Lots
Description: Geometric mean titer (GMT) of RSV A and RSV B neutralizing antibodies were calculated by exponentiating the mean logarithm of the titers and the corresponding 95% confidence interval (CI) was based on the Student t distribution. GMTs were reported in the descriptive section. Geometric mean ratios (GMRs) for each RSV vaccine lot comparison (Group 1/Group 2, Group 1/Group 3, and Group 2/Group 3) for RSV A and RSV B neutralizing antibody titers was calculated and reported in statistical analysis.
Time Frame: 1 month (27 to 42 days window) after vaccination on Day 1
Population: Evaluable immunogenicity population included all eligible participants who received vaccine to which they were randomized at visit 1, had a valid and determinate immunogenicity result from the blood sample collected within 27 to 42 days after vaccination and had no other major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: RSVpreF Lot 1 | Group 2: RSVpreF Lot 2 | Group 3: RSVpreF Lot 3
Number analyzed (Participants) | 236 | 236 | 238
Titer
  RSV A | 25238.1 [22867.7 to 27854.2] | 25207.5 [22360.8 to 28416.6] | 24130.9 [21536.3 to 27038.1]
  RSV B | 21701.9 [19433.1 to 24235.6] | 20317.3 [17944.4 to 23003.9] | 19238.1 [16920.0 to 21873.9]
Statistical Analysis 1: Comparison: Group 1: RSVpreF Lot 1 vs Group 2: RSVpreF Lot 2; RSV A; Test type: Equivalence — Equivalence was established if the 2-sided 95% CI for the ratio of neutralizing GMTs for each pair of individual vaccine lots (RSVpreF Lot 1/RSVpreF Lot 2, RSVpreF Lot 1/RSVpreF Lot 3 and RSVpreF Lot 2/RSVpreF Lot 3) was within the interval (0.667, 1.5), for both antigens simultaneously; Geometric Mean Ratio = 1.00, 95% CI 2-sided [0.858 to 1.169] — GMRs and 2-sided CIs were calculated by exponentiating the difference in least-square (LS) means and corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model
Statistical Analysis 2: Comparison: Group 1: RSVpreF Lot 1 vs Group 3: RSVpreF Lot 3; RSV A; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.05, 95% CI 2-sided [0.900 to 1.215] — GMRs and 2-sided CIs were calculated by exponentiating the difference in LS means and corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model
Statistical Analysis 3: Comparison: Group 2: RSVpreF Lot 2 vs Group 3: RSVpreF Lot 3; RSV A; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.04, 95% CI 2-sided [0.886 to 1.232] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Group 1: RSVpreF Lot 1 vs Group 2: RSVpreF Lot 2; RSV B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.07, 95% CI 2-sided [0.905 to 1.261] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Group 1: RSVpreF Lot 1 vs Group 3: RSVpreF Lot 3; RSV B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.13, 95% CI 2-sided [0.953 to 1.336] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Group 2: RSVpreF Lot 2 vs Group 3: RSVpreF Lot 3; RSV B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.06, 95% CI 2-sided [0.884 to 1.262] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination
Description: Local reactions included pain at injection site, redness and swelling and were recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm) and graded as mild: greater than (>) 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with activity, moderate: interfered with activity and severe: prevented daily activity. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after vaccination on Day 1
Population: Safety population included all randomized participants who received study intervention. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Data for this outcome measure was planned to be analyzed for placebo and pooled RSVpreF lots (Groups 1, 2, and 3).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RSVpreF Pooled Lots (Groups 1, 2 and 3): Participants were randomized to receive a single intramuscular injection of 120 mcg RSVpreF lots 1, 2 or 3 reconstituted with sterile water for injection, once only on Day 1.
Arm/Group | Placebo | RSVpreF Pooled Lots (Groups 1, 2 and 3)
Number analyzed (Participants) | 247 | 742
Percentage of participants
  Pain at injection site: Mild | 10.5 [7.0 to 15.0] | 31.5 [28.2 to 35.0]
  Pain at injection site: Moderate | 0.8 [0.1 to 2.9] | 5.4 [3.9 to 7.3]
  Pain at injection site: Severe | 0 [0.0 to 1.5] | 0 [0.0 to 0.5]
  Redness: Mild | 0.4 [0.0 to 2.2] | 4.4 [3.1 to 6.2]
  Redness: Moderate | 0.4 [0.0 to 2.2] | 2.8 [1.8 to 4.3]
  Redness: Severe | 0 [0.0 to 1.5] | 0.5 [0.1 to 1.4]
  Swelling: Mild | 0.4 [0.0 to 2.2] | 4.0 [2.7 to 5.7]
  Swelling: Moderate | 0 [0.0 to 1.5] | 3.8 [2.5 to 5.4]
  Swelling: Severe | 0 [0.0 to 1.5] | 0 [0.0 to 0.5]

3. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and were recorded by participants in an e-diary. Fever was defined as temperature greater than or equal to (>=)38.0 degrees Celsius (C) and categorized as mild (>=38.0 to 38.4 degrees C), moderate (>38.4 to 38.9 degrees C) and severe (>38.9 to 40.0 degrees C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours (h), moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after vaccination on Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | RSVpreF Pooled Lots (Groups 1, 2 and 3)
Number analyzed (Participants) | 247 | 742
Percentage of participants
  Fever: Mild | 0.4 [0.0 to 2.2] | 0.8 [0.3 to 1.8]
  Fever: Moderate | 0.4 [0.0 to 2.2] | 0.9 [0.4 to 1.9]
  Fever: Severe | 0 [0.0 to 1.5] | 0.3 [0.0 to 1.0]
  Fatigue: Mild | 19.4 [14.7 to 24.9] | 21.3 [18.4 to 24.4]
  Fatigue: Moderate | 12.6 [8.7 to 17.3] | 21.0 [18.1 to 24.1]
  Fatigue: Severe | 1.2 [0.3 to 3.5] | 0.4 [0.1 to 1.2]
  Headache: Mild | 18.2 [13.6 to 23.6] | 21.3 [18.4 to 24.4]
  Headache: Moderate | 10.1 [6.7 to 14.6] | 14.8 [12.3 to 17.6]
  Headache: Severe | 0 [0.0 to 1.5] | 0.1 [0.0 to 0.7]
  Nausea: Mild | 4.5 [2.2 to 7.8] | 6.3 [4.7 to 8.3]
  Nausea: Moderate | 2.4 [0.9 to 5.2] | 4.2 [2.9 to 5.9]
  Nausea: Severe | 0 [0.0 to 1.5] | 0 [0.0 to 0.5]
  Vomiting: Mild | 0.4 [0.0 to 2.2] | 1.1 [0.5 to 2.1]
  Vomiting: Moderate | 0 [0.0 to 1.5] | 0.5 [0.1 to 1.4]
  Vomiting: Severe | 0 [0.0 to 1.5] | 0 [0.0 to 0.5]
  Diarrhea: Mild | 5.7 [3.1 to 9.3] | 8.9 [6.9 to 11.2]
  Diarrhea: Moderate | 4.9 [2.5 to 8.3] | 4.2 [2.9 to 5.9]
  Diarrhea: Severe | 0.4 [0.0 to 2.2] | 0.4 [0.1 to 1.2]
  Muscle Pain: Mild | 7.7 [4.7 to 11.8] | 17.3 [14.6 to 20.2]
  Muscle Pain: Moderate | 3.2 [1.4 to 6.3] | 12.3 [10.0 to 14.8]
  Muscle Pain: Severe | 0 [0.0 to 1.5] | 0.1 [0.0 to 0.7]
  Joint Pain: Mild | 2.8 [1.1 to 5.8] | 8.2 [6.3 to 10.4]
  Joint Pain: Moderate | 1.6 [0.4 to 4.1] | 6.7 [5.0 to 8.8]
  Joint Pain: Severe | 0 [0.0 to 1.5] | 0 [0.0 to 0.5]

4. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs included both serious and all non-serious adverse events excluding local reactions and systemic events. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; required inpatient hospitalization or prolongation of existing hospitalization; life-threatening ; persistent or significant disability/incapacity; congenital anomaly/birth defect and suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Day of consent (Day 1) through study completion (approximately 1 Month)
Population: Safety population included all randomized participants who received study intervention. Data for this outcome measure was planned to be analyzed for placebo and pooled RSVpreF lots (Groups 1, 2, and 3).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | RSVpreF Pooled Lots (Groups 1, 2 and 3)
Number analyzed (Participants) | 247 | 745
Percentage of participants
  AE | 6.1 [3.4 to 9.8] | 5.8 [4.2 to 7.7]
  SAE | 0 [0.0 to 1.5] | 0 [0.0 to 0.5]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events (systematic assessment): within 7 days after vaccination on Day 1; AEs and SAEs (non-systematic assessment) and all-cause mortality: Day of consent (Day 1) through study completion (approximately 1 Month)
Description: Safety population included all randomized participants who received study intervention.
Arm/Group | Placebo | Group 1: RSVpreF Lot 1 | Group 2: RSVpreF Lot 2 | Group 3: RSVpreF Lot 3 | RSVpreF Pooled Lots (Groups 1, 2 and 3)
All-Cause Mortality (participants affected / at risk) | 0/247 | 0/249 | 0/247 | 0/249 | 0/745
Serious Adverse Events (participants affected / at risk) | 0/247 | 0/249 | 0/247 | 0/249 | 0/745
Other Adverse Events (participants affected / at risk) | 130/247 | 170/249 | 172/247 | 166/249 | 508/745
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=247) | Group 1: RSVpreF Lot 1 (N=249) | Group 2: RSVpreF Lot 2 (N=247) | Group 3: RSVpreF Lot 3 (N=249) | RSVpreF Pooled Lots (Groups 1, 2 and 3) (N=745)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3 | 5
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 27 | 35 | 38 | 27 | 100
Nausea (NAUSEA) (Gastrointestinal disorders) | 17 | 23 | 29 | 26 | 78
Vomiting (VOMITING) (Gastrointestinal disorders) | 1 | 3 | 5 | 4 | 12
Axillary pain (General disorders) | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 2 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 2
Fatigue (FATIGUE) (General disorders) | 82 | 107 | 103 | 107 | 317
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 1
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 28 | 83 | 97 | 94 | 274
Injection site rash (General disorders) | 0 | 0 | 1 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (FEVER) (General disorders) | 2 | 4 | 7 | 4 | 15
Swelling (General disorders) | 0 | 0 | 1 | 0 | 1
Swelling (SWELLING) (General disorders) | 1 | 11 | 23 | 24 | 58
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 0 | 2 | 4
Ear infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 4 | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 1
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 11 | 37 | 35 | 39 | 111
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 27 | 68 | 82 | 70 | 220
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Headache (HEADACHE) (Nervous system disorders) | 70 | 95 | 88 | 86 | 269
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 2 | 11 | 23 | 24 | 58
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT05096208/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT05096208/SAP_001.pdf